CLINICAL TRIAL: NCT05684562
Title: Pulmonary Determinants of Cardiorespiratory Fitness in Patients With Fontan Procedure
Brief Title: Pulmonary Determinants of Cardiorespiratory Fitness in Fontan Patients
Status: Recruiting | Type: Observational
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Haluk TEKERLEK, Research assistant, Hacettepe University
Other Study IDs: fontanpulmonarydeterminants
Record Dates: First submitted 2022-12-27; First posted 2023-01-13 (Actual); Last update posted 2024-03-28 (Actual); Status verified 2024-03

CONDITIONS: Fontan Procedure; Congenital Heart Disease
MeSH Terms: conditions — Heart Defects, Congenital | interventions — Exercise Test; Respiratory Physiological Phenomena

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Fontan group: Cardiopulmonary exercise test Pulmonary function test respiratory muscle strength test
  Interventions: Other: Cardiopulmonary exercise test; Other: Pulmonary function test; Other: Respiratory muscle strength test
- Control Group: Cardiopulmonary exercise test Pulmonary function test respiratory muscle strength test
  Interventions: Other: Cardiopulmonary exercise test; Other: Pulmonary function test; Other: Respiratory muscle strength test

INTERVENTIONS:
Other: Cardiopulmonary exercise test — CPET, the gold standard, will be used in the assessment of cardiorespiratory fitness. The cardiopulmonary exercise test system (Cosmed Quark CPET, Rome, Italy) is a safe method in which the patient can be monitored via ECG during the execution of the individual on a treadmill, and simultaneously lactate measurement, maximal O2 consumption, and CO2 production are evaluated. The Bruce protocol is the most commonly used method for KPET applied with a treadmill. However, since the Bruce protocol prefers high workload preferences, the Modified Bruce/half Bruce protocol with intermediate increments will be used. In addition, dyspnea, leg fatigue, and general fatigue at rest, during the test, and during the recovery phases after the test will be recorded with a sphygmomanometer using the Modified Borg Scale.
Other: Pulmonary function test — Pulmonary function testing will be performed with a spirometer (Cosmed Quark CPET, Rome, Italy) connected to the CPET system using standard procedures. Forced vital capacity (FVC), forced expiratory volume in 1 second (FEV1), FEV1/FVC, peak expiratory volume measured at 25% and 75% of forced expiratory time (FEF 25-75%), and peak expiratory volume (PEF) parameters will be saved.
Other: Respiratory muscle strength test — Intraoral maximum inspiratory pressure (MIP) and maximum expiratory pressure (MEP) will be used as indicators of respiratory muscle strength. A portable intraoral pressure gauge (MicroRPM, Micromedical, Kent, UK) and nose clip will be used during MIP and MEP assessments. MIP and MEP measurements will be obtained using standard procedures. 3 measurements will be made where the difference between each measurement is not more than 10% and the maximum value of MIP and MEP will be recorded.

SUMMARY:
This study will examine and record the patient's medical information and medical records (patient files, computer records, etc.). Physical examination, echocardiographic, electrocardiographic, laboratory, radiological, etc. evaluations are made during the routine controls of the patients. Within the scope of this study, no attempt will be made on the patients, no additional tests will be performed, or treatment changes will not be made in the patients because they are included in this study. After these records, KPET will be performed by a specialist doctor and physiotherapist for the patients who are directed to the Faculty of Physical Therapy and Rehabilitation Cardiopulmonary Rehabilitation Unit. Pulmonary function tests and respiratory muscle strength measurements will be performed on patients who have adequate rest after CPET.

ELIGIBILITY:
Fontan Group Inclusion Criteria:

* Be between 8-55 years old
* Having undergone a Fontan operation
* Clinical stability of the patients (preserved ventricular function)
* No change in ongoing drug therapy that adversely affects clinical stability
* At least 1 year after the operation

Fontan Group Exclusion Criteria:

* Neurological and/or genetic musculoskeletal disease
* Having orthopedic and cognitive problems that prevent testing
* The patient's and/or family's unwillingness to participate in the study

Control Group Inclusion Criteria:

* Not have cardiovascular, neurological, and/or genetic musculoskeletal disease
* Not having orthopedic and cognitive problems that prevent testing
* The patient's and/or family's willingness to participate in the study

Ages: 8 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Patients aged 8-55 years who underwent the Fontan procedure and followed up by Department of Pediatric Cardiology will be included in the study. In the evaluation of patients in terms of suitability for the study, a detailed history, medical and family history, and a physical examination focused on all systems. The eligible patients will be referred to the Cardiopulmonary Rehabilitation Unit after the routine evaluations including demographic and clinical characteristics and laboratory tests are completed. For patients aged 8-17 years, the parental informed consent form for the research study and the child consent form for the research study will be carefully explained and included in the study after the parents and patients have read, understood, and accepted. For patients aged 18 years and older, the informed consent form for the research study will be carefully explained and will be included in the study after the patients have read, understood, and accepted.
Sampling Method: Non-Probability Sample
Enrollment: 78 (Estimated)
Dates: Start 2023-12-26 (Actual); Primary Completion 2024-12-25 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Maximal oxygen consumption | 30-45 minutes
Forced vital capacity (FVC) | 15-20 minutes
Forced expiratory volume in 1 second (FEV1) | 15-20 minutes
FEV1/FVC | 15-20 minutes
Maximal inspiratory pressure | 15-20 minutes
Maximal expiratory pressure | 15-20 minutes
Ratio curve of minute ventilation to carbon dioxide production (VE/VCO2) slope | 30-45 minutes
Ratio of minute ventilation to carbon dioxide production (VE/VCO2) | 30-45 minutes
Oxygen uptake efficiency slope (OUES) | 30-45 minutes
Minute ventilation (VE) | 30-45 minutes
End tidal oxygen pressure (PetO2) | 30-45 minutes
End tidal carbon dioxide pressure (PetCO2) | 30-45 minutes

CONTACTS AND LOCATIONS:
Locations (1):
- Hacettepe Unıversity, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No